CLINICAL TRIAL: NCT01553630
Title: Reamed Locked Plating - Metaphyseal Fractures of the Distal Femur and Tibia
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Low enrollment.
Sponsor: Florida Orthopaedic Institute (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: Reamed Locked Plating
Record Dates: First submitted 2012-03-08; First posted 2012-03-14 (Estimated); Last update posted 2014-11-11 (Estimated); Status verified 2014-11

CONDITIONS: Femoral Fractures; Tibial Fractures
Keywords: Fractures; distal femur fractures; distal tibial fracures
MeSH Terms: conditions — Femoral Fractures; Tibial Fractures; Fractures, Bone; Femoral Fractures, Distal | interventions — Surgical Procedures, Operative; Bone Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- RIA bone graft (Active Comparator): Surgery: open reduction and internal fixation (ORIF) of high energy metaphyseal fractures with Reamed Irrigator Aspirator (RIA) bone graft at the time of fixation.
  Interventions: Procedure: RIA bone graft
- Surgery without bone graft (Active Comparator): Surgery:open reduction and internal fixation (ORIF) of high energy metaphyseal fractures without Reamed Irrigator Aspirator (RIA) bone graft at the time of fixation.
  Interventions: Procedure: Surgery without bone graft

INTERVENTIONS:
Procedure: RIA bone graft — Acute autogenous bone grafting with RIA graft at the time of surgical fixation.
  Arms: RIA bone graft
Procedure: Surgery without bone graft — Plating of fracture without bone graft
  Arms: Surgery without bone graft

SUMMARY:
Comminuted metaphyseal fractures (OTA classification A2/3 and C2/3) of the distal femur and distal tibia are difficult to treat and typically have more complications than other metaphyseal fractures. Delayed union, nonunion and need for secondary bone graft procedures are frequent outcomes. These A2/3 and C2/3 fractures of the distal femur and distal tibia treated with locked plates often have a critical sized fracture gap (poorly organized cortical pieces many of which are stripped of soft tissue). Optimal management strategies that minimize both fracture healing time and complication rates remain controversial. Primary bone grafts or early secondary bone grafts have been recommended for these comminuted open fractures, but have not been studied as the primary end point in a randomized trial. There is a need to study primary bone grafting during open reduction and internal fixation (plating) of these difficult fractures, to determine if shorter healing time, and thus less need for reoperation, can be achieved.

Hypothesis Acute autogenous bone grafting at the time of fixation will hasten clinical and radiographic union with a lower need for secondary procedures

DETAILED DESCRIPTION:
Study procedures:

Eligible fractures will be identified, consented and randomized to RIA augmentation or non graft treatment. Bone graft will be harvested through the fracture at the time of the definitive fixation procedure. No additional graft can be utilized acutely (No iliac crest bone graft, or INFUSE, OP-1, Callos, etc).

Randomization Procedures: We will be using Research Randomizer to calculate a random assignment design for Group A and Group B, which will be kept by the Research Coordinator. Once a patient agrees to participate in the study and signs an Informed Consent Form, the treating surgeon will request the treatment assignment from the Research Coordinator prior to the surgery. Group A will receive RIA augmentation. Group B will receive non-graft treatment. Patient outcomes will be analyzed using intention to treat principles.

Surgical Procedures: Locked lateral plating of comminuted supracondylar femur and distal tibia fractures is an accepted standard of care. In severely comminuted fracture patterns, restoration of length and alignment often leaves substantial fracture gap increasing the risk of fracture nonunion. Historically, this has been accepted with the plan to return to the patient to surgery for bone grafting at a later date if the nonunion is developing. Intra-focal reaming with irrigation & aspiration (RIA) at time of initial surgery allows for acute autogenous bone grafting with no increased morbidity to the patient.

Surgery for Group A receiving bone graft follows the same course as without acute grafting (same incision, dissection etc.) with the exception that after initial exposure, a guide wire is placed into the proximal femoral canal (retrograde) through the fracture, and graft is harvested using the RIA system. The RIA system has a reservoir to collect the reamings as they are aspirated from the fracture site. Reduction and fixation with locked plates then proceed as usual and the harvested graft is then placed into the residual gap with the expectation that nonunion rates may be decreased. A theoretical advantage is the renewed fracture hematoma that will collect at the fracture site secondary to reaming the canal which may also increase union rates and time to union. No increased morbidity is incurred and the increased surgical time is under 10 minutes.

ELIGIBILITY:
Inclusion Criteria:

* High energy metaphyseal fracture (distal femur or tibia) indicated for plate fixation (open or closed)
* Adult, acute fractures only

Exclusion Criteria:

* Unable to ream fractured bone
* Subject is unable, unwilling or unlikely to follow up
* Subject is under age 18 years
* Prisoners

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2010-05; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Time to union | 3 months, 6 months and 1 year
  This will be evaluated with the reading of xrays

SECONDARY OUTCOMES:
Reoperation rate | 3 months, 6 months, 1 year
  The rate of re operation will be evaluated

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Tampa General Hospital, Tampa, Florida
  - St Jospehs Hospital, Tampa, Florida

REFERENCES:
- [Derived] Claireaux HA, Searle HKC, Parsons NR, Griffin XL. Interventions for treating fractures of the distal femur in adults. Cochrane Database Syst Rev. 2022 Oct 5;10(10):CD010606. doi: 10.1002/14651858.CD010606.pub3. PMID 36197809